CLINICAL TRIAL: NCT06252441
Title: Comparative Clinical Study to Evaluate the Possible Efficacy and Safety of Oral N-Acetyl Cysteine Versus Rectal Diclofenac in the Prevention of Post Endoscopic Retrograde Cholangiopancreatography Pancreatitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mariam Tarek Mohammed Tabana, Teaching Assistant , Faculty of Pharmacy, Menoufia University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Post ERCP Pancreatitis
Record Dates: First submitted 2024-01-31; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Post ERCP Pancreatitis
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectal Diclofenac (Active Comparator): This Group will include 23 patients who will receive 100 mg rectal diclofenac before ERCP.
  Interventions: Drug: Rectal Diclofenac
- Oral N-acetyl cysteine (Active Comparator): This Group will include 23 patients who will receive 1200 mg N-acetyl cysteine in 150 cc water orally before ERCP.
  Interventions: Drug: Oral N-acetyl cysteine

INTERVENTIONS:
Drug: Rectal Diclofenac — 100 mg Rectal Diclofenac Before ERCP
  Arms: Rectal Diclofenac
Drug: Oral N-acetyl cysteine — 1200 mg N-acetyl cysteine in 150 cc water orally before ERCP.
  Arms: Oral N-acetyl cysteine

SUMMARY:
The aim of the current study is to compare the efficacy and safety of oral NAC and rectal diclofenac in preventing Post Endoscopic retrograde cholangiopancreatography Pancreatitis. .

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) , a key tool that is used in diagnosis and treatment of pancreato-biliary diseases. Post-ERCP pancreatitis (PEP) is the most common and serious complication that can occur following this procedure and can lead to significant morbidity and mortality. A variety of patient-related and procedure-related factors have been associated with higher rates of PEP.

Two definitions were used for diagnosis of PEP. In both definitions, PEP is diagnosed if two of the three criteria are found in the patient .The consensus criteria that was developed by Cotton and Colleagues in 1991 defined PEP as the presence of a new pancreatic-type abdominal pain associated with at least a threefold elevation in pancreatic enzyme concentration occurring 24 hours following the ERCP procedure, with the necessity for a new or extended hospitalization for at least two nights. Severity of pancreatitis is defined based on the number of hospitalized days following ERCP as mild (< 4 days), moderate (4 to 10 days), or severe (>10 days). The revised Atlanta Classification in 2012 lists abdominal pain consistent with acute pancreatitis, amylase or lipase elevation to more than 3 times the upper limit of normal, and abdominal imaging that reveals pancreatic inflammation.

Several potential triggers can contribute to PEP. Mechanical trauma caused by ERCP instrumentation can harm the papilla and pancreatic duct, affecting pancreatic drainage. Thermal injury can occur during biliary or pancreatic sphincterotomy electrosurgical current. Chemical damage can occur when contrast medium is introduced into the pancreatic duct. Hydrostatic damage can occur when injecting contrast media into the pancreatic duct or infusing fluids such as water or saline solution during sphincter manometry. Regardless of the cause, the initial injury sets in motion a chain of events that include premature activation of proteolytic enzymes, autodigestion of pancreatic tissue, and impaired secretion from acinar cells. These events result in pancreatitis clinical symptoms, which have an influence both locally and systemically. Most PEP prevention techniques try to disrupt one or more steps in this cascade.

While the precise mechanism of PEP remains unknown, it is most likely induced by a proinflammatory cascade initiated by pancreatic acinar cell damage, which results in systemic cytokine release. Cytokines play a major role in the pathogenesis of acute pancreatitis as part of the underlying systemic inflammatory response, tissue damage, and organ dysfunction. Tumor necrosis factor alpha (TNF-α) is a pro-inflammatory cytokine that promotes the inflammatory response, whereas Interleukin-10 (IL-10) is an immunosuppressive cytokine that inhibits inflammation. These markers can be used in measurement of the degree of systemic inflammation as predictors of the development of PEP.

Phospholipase A2 is essential in this signaling cascade. Diclofenac is a nonsteroidal anti-inflammatory drug (NSAID) that effectively inhibits phospholipase A2 activity. According to this notion, anti-inflammatory drugs such as diclofenac can stop or attenuate the first cascade that leads to clinical PEP.

Previous meta-analyses have suggested that NSAIDs are effective in preventing PEP. The European Society of Gastrointestinal Endoscopy guidelines recommend routine rectal administration of 100 mg of diclofenac or indomethacin immediately before ERCP procedure in all patients without contraindications to NSAIDs administration. Rectal administration route of diclofenac is the most effective in the prevention of PEP. Rectal diclofenac is a cheap, widely available agent with easy administration method and favorable side effect profile.

Oxidative stress and active oxygen species can activate inflammatory cascade and immune responses. N-acetyl cysteine (NAC), an antioxidant drug with anti-inflammatory properties can inhibit oxidative stress as well as inflammatory intermediates, suggesting that it could aid in the prevention of PEP. Despite the failure of intravenous N-acetyl cysteine studies, 2013 pilot research revealed that oral NAC may be useful in reducing PEP. This would be due to the different pharmacokinetics of NAC followed in different studies. In a multicenter global randomized controlled trial investigation, It is reported that oral NAC is more effective than indomethacin in the prevention of PEP.

Although both oral NAC and rectal diclofenac are widely used pharmacological agents, till now no study has evaluated their comparative safety and efficacy in preventing PEP. Hence this study is planned to evaluate and compare their efficacy and safety in preventing PEP.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years old.
2. Gender: males and females.
3. Patients with suitable indications for ERCP due to suspected pancreato-biliary disorders.
4. Blood amylase and lipase levels before ERCP are within the normal limits.

Exclusion Criteria:

1. Age of less than 18 years old.
2. Uncontrolled diabetes mellitus (DM).
3. Severe bleeding tendency.
4. Impaired renal function (serum creatinine > 2 mg/dL), (creatinine clearance <30 ml/min).
5. Patients with severe heart disease.
6. Subjects who underwent prior biliary or pancreatic sphincterotomy or dilatation or stenting of either duct.
7. Currently pregnant or nursing.
8. Admission due to established pancreatitis before ECRP.
9. Unwillingness to undergo ERCP.
10. Previously documented allergy to NAC or diclofenac or any other NSAIDs.
11. History of NSAIDs intake one week before the procedure.
12. Recent Active bleeding, ulcer, or asthma.
13. Patients with rectal disease (hemorrhoids, fissures, abscesses, and incontinence).

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The development of pancreatitis after the procedure according to consensus criteria | Before performing ERCP, baseline serum amylase and lipase levels will be measured in all patients. After twenty four ( 24) hours post ERCP procedure, patients' serum amylase and lipase levels will be measured.
  Briefly in this criteria PEP will be diagnosed if the patient met two of the three following criteria after ERCP:
  A- New onset or increased abdominal pain consistent with acute pancreatitis B- Pancreatic enzyme elevation to at least three times the upper limit of normal at twenty four (24) hours after the procedure C- Necessity for new or continued hospitalization for at least two nights
The change in the serum levels of Tumor necrosis factor alpha (TNF-α) and Interleukin-10 (IL-10 )before and after ERCP procedure | Biomarkers will be measured at baseline before the ERCP procedure and twenty four (24 ) hours after the procedure
  These markers measure the degree of systemic inflammation as predictors of the development of PEP.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstructive Jaundice Clinic in the National Liver Institute, Menoufia University , Shebin Elkoom, Menofia, Egypt

IPD SHARING:
Plan to Share IPD: No